CLINICAL TRIAL: NCT03568409
Title: Efficacy of ABO-GLYC on Glycemic and Metabolic Status of Patients With Type 2 Diabetes
Brief Title: ABO-GLYC in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: Latis S.r.l. (Industry); Fondazione Edmund Mach (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABO-GLYC-16
Record Dates: First submitted 2018-05-15; First posted 2018-06-26 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2021-07

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: ABO-GLYC (Experimental): Libramed
  Interventions: Device: ABO-GLYC
- Group B: Placebo (Placebo Comparator)
  Interventions: Other: ABO-GLYC Placebo

INTERVENTIONS:
Device: ABO-GLYC — 3 tablets twice a day, before the main meals (lunch and dinner) continuatively for 24 weeks.
  Other Names: Libramed
  Arms: Group A: ABO-GLYC
Other: ABO-GLYC Placebo — 3 tablets twice a day, before the main meals (lunch and dinner) continuatively for 24 weeks.
  Arms: Group B: Placebo

SUMMARY:
Evaluation of the improvement of the overall glycemic control after 6 months of treatment with ABO-GLYC, as a result of reduction of HbA1c and/or post-prandial glycemic peak.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with diagnosis of type 2 diabetes, aged 18-75
2. HbA1c at screening between 6.5% and 7.5%
3. Last 2 HbA1c values in the last 12 months between 6.5% and 7.5%
4. Intolerance to metformin without unquestionable indication to other oral hypoglycemic agents
5. BMI 25-38 kg/m2
6. Willing and able to understand and sign the informed consent and complete the patient diary provided
7. Women participant of childbearing age should be negative to pregnancy test (performed on blood), and will have to use an appropriate contraceptive method throughout the study.

Exclusion Criteria:

1. Micro and macrovascular complication of diabetes in advanced stage (i.e., proliferative diabetic retinopathy; chronic renal failure III-IV stage KDOQI)
2. Chronic gastro-intestinal disease
3. Heavy smoker subjects
4. Alcohol abuse
5. Chronic liver and kidney disease (AST or ALT values > 2.5 UNL or plasma creatinine > 1.5 mg/dl)
6. Previous major gastrointestinal surgery
7. History of eating disorders
8. Pregnancy or lactation
9. Use of food supplements containing in particular but not limited to fibers and polysaccharides, in the last six months with frequency and dosage such as to interfere with the study.
10. Autoimmune diseases
11. Known hypersensitivity to any of the components of the product.
12. Any condition which prevent subject participation in the opinion of the principal investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of the overall glycemic control after 6 months of treatment with ABO-GLYC, as a result of reduction of HbA1c and/or post-prandial glycemic peak. | Week0 and Week24
  HbA1c measure
Improvement of the overall glycemic control after 6 months of treatment with ABO-GLYC, as a result of reduction of HbA1c and/or post-prandial glycemic peak. | Week0 and Week24
  Tmax
Improvement of the overall glycemic control after 6 months of treatment with ABO-GLYC, as a result of reduction of HbA1c and/or post-prandial glycemic peak. | Week0 and Week24
  Cmax

SECONDARY OUTCOMES:
Improvement of markers of glycemic variability (plasma glucose level) | Week0 to Week24
  Composite measurement of standard deviation and coefficient of variation of the plasma glucose level
Improvement of markers of glycemic variability (MAGE) | Week0 to Week24
  mean amplitude of glucose excursion (MAGE)
Improvement of markers of glycemic variability (HBGl) | Week0 to Week24
  high blood glycemic index (HBGI)
Improvement of markers of glycemic variability (LBGI) | Week0 to Week24
  , low blood glycemic index (LBGI)
Improvement of markers of glycemic variability (hypo/hyper glycemia) | Week0 to Week24
  percentage of time spent in hypoglycemia or hyperglycemia
Improvement of markers of metabolic status (BMI) | Week0 to Week24
  Weight and height will be combined to report BMI in kg/m^2,total cholesterol, LDL triglycerides or NEFA, HDL and in the percentage of body fat determined by bioimpedentiometry
Improvement of markers of glyco-oxidative stress | Week0 to Week24
  Measurement of receptor for advanced glycation endproducts (RAGE), Malondialdehyde (MDA) and/or oxidized LDL
Improvement of markers of inflammation | Week0 to Week24
  Measurement of TNF-alpha, IL-1, IL-6
Improvement of markers of metabolic status (lipid profile) | Week0 to Week24
  Measurement of total cholesterol, HDL cholesterol and Tryglycerides
Improvement of markers of metabolic status (body composition) | Week0 to Week24
  percentage of body fat determined by bioimpedentiometry
Evaluation of gut microbiome changes (bacteria population) | Week 0, Week 1, Week 12, Week 24
  Evaluation of bacteria population
Evaluation of gut microbiome changes (SCFA) | Week 0, Week 1, Week 12, Week 24
  Evaluation of short change fatty acids measurements (SCFA)
Improvement in markers of insulin resistance | Week 0 and Week 24
  Measurement of HOMA-IR and QUICKI
Improvement in markers of insulin secretion after standardized meal. | Week 0 and Week 24
  Measurement of insulin and c-peptide secretion measured during the glycemic curve after a standardized meal
Evaluation of the dietary adherence | Week0 to Week24
  Perceived Dietary Adherence Questionnaire (PDAQ). The PDAQ uses a 5-point Likert scale to assess perceived difficulty.
Adverse events (AEs) evaluation and product tolerability. | Week0 to Week24
  Adverse event will be recorded during the course of the study, after the signature of the informed consent
Control of the glycemia. | Week0 to Week24
  The data from the glycemic diary will be monitored to assess the good control of the glycemia as measured by Self Monitoring of Blood Glucose (SMBG).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No